CLINICAL TRIAL: NCT06337123
Title: A Post Market Clinical Study Evaluating Clinical and Radiographic Outcomes of Total Knee Arthroplasty With Physica Porous KR or Physica Porous PS in Combination With Physica TT Tibial Plate in Cementless Configuration.
Brief Title: Physica TT Tibial Plate Follow up Study
Status: Recruiting | Type: Observational
Sponsor: Limacorporate S.p.a (Industry)
Responsible Party: Sponsor
Other Study IDs: K-38
Record Dates: First submitted 2024-03-15; First posted 2024-03-29 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Knee Arthropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Physica Porous KR femoral component: Devices: Physica TT Tibial Plate and Physica Porous KR femoral component
  Total knee arthroplasty with Physica TT Tibial Plate and Physica Porous KR femoral component
  Interventions: Device: Device: Physica TT TIbial Plate and Physica Porous KR
- Physica Porous PS femoral component: Devices: Physica TT Tibial Plate and Physica Porous PS femoral component
  Total knee arthroplasty with Physica TT Tibial Plate and physica Porous PS femoral component
  Interventions: Device: Device: Physica TT TIbial Plate and Physica Porous PS

INTERVENTIONS:
Device: Device: Physica TT TIbial Plate and Physica Porous KR — Devices: Physica TT Tibial Plate and Physica Porous KR femoral component
  Data collection of population that underwent total knee arthroplasty with Physica TT Tibial Plate and Physica Porous KR femoral component
  Groups: Physica Porous KR femoral component
Device: Device: Physica TT TIbial Plate and Physica Porous PS — Devices: Physica TT Tibial Plate and Physica Porous KR femoral component
  Data collection of population that underwent total knee arthroplasty with Physica TT Tibial Plate and Physica Porous PS femoral component
  Groups: Physica Porous PS femoral component

SUMMARY:
This clinical study aims at evaluating clinical, radiographic, patient-reported outcomes of total knee arthroplasty with Physica TT Tibial Plate in combination with Physica Porous KR or Physica Porous PS up to 2 years after surgery, in order to assess the performance of the devices. Furthermore, ithe objective is to collect short-term survivorship of the implant and the incidence of early complications.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female of any race requiring a total knee replacement (TKR) and suitable for receiving Physica Porous KR or Physica Porous PS femoral component in combination with Physica TT Tibial Plate.
2. Age ≥ 18 years old.
3. Candidate for primary total knee replacement when clinical indications based on physical examination and medical history include one or more of the following conditions:

   1. Non-inflammatory degenerative joint disease like knee osteoarthritis, post traumatic knee arthritis
   2. Inflammatory degenerative joint disease like rheumatoid arthritis
   3. Any other medical reason for which the investigator deems the subject as a possible candidate for total knee replacement.
4. Patient has well-preserved and well-functioning collateral ligaments and one of the following conditions:

   1. Absent or not-functioning posterior cruciate ligament and severe antero-posterior instability of the knee joint (for Physica Porous PS)
   2. Undamaged and functional posterior cruciate ligament (for Physica Porous KR)
5. Patient is able to understand the conditions of the study, to comply with the prescribed rehabilitation as well as willing to perform all scheduled follow-up visits.
6. Patient signed the study-specific informed consent form approved by the ethics committee before study activities

Exclusion Criteria:

1. Severe instability of the knee joint secondary to the absence of collateral ligament integrity and/or function. Only for Physica Porous KR: important joint instability and deficiency of posterior cruciate ligament.
2. Any active or suspected infection (local or systemic) or previous history of infection that may affect the prosthetic joint.
3. Previous partial knee replacement (unicompartmental, bicompartmental or patellofemoral joint replacement), patellectomy, high tibial osteotomy.
4. Significant bone loss on femoral or tibial joint side.
5. Affected by malignant cancer with life expectancy less than 2 years or where cancer treatment might affect the normal postoperative course.
6. Known incompatibility or allergy to the product materials, and/or metal hypersensitivity to implant materials.
7. Septicaemia.
8. Persistent acute or chronic osteomyelitis.
9. Open epiphyses (immature patient with active bone growth).
10. Necrotic bone
11. Arterial vascular insufficiency or nerve diseases of the lower limbs severe enough to interfere with the study evaluation.
12. Compromised bone stock due to disease, infection or prior implantation that cannot provide adequate support and/or fixation to the prosthesis.
13. Systemic or metabolic disorders leading to progressive bone deterioration, which may impair fixation and stability of the implant.
14. Any concomitant disease and dependency that might affect the performance of the implanted prosthesis.
15. Any clinically major pathology based on clinical medical history or any medical intervention or reason that the Investigator feels may affect the study evaluation.
16. Neurological or musculoskeletal disorder or disease that may adversely affect gait, functional recovery and evaluation.
17. Neuromuscular or neurosensory deficit that would hamper the performance assessment of the device.
18. Any psychiatric illness that would prevent comprehension of the details and nature of the study.
19. Simultaneously taking part in another surgical intervention study or pain management study that may affect with clinical study outcomes.
20. Female patient who is pregnant, nursing, or planning a pregnancy.
21. Important osteoporosis, haemophilic disease.
22. Internistic problems with high risk for surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General population of subjects requiring a primary TKR with a diagnosis of painful primary or secondary osteoartrithis not responding to other conservative treatments, after the review of medical history and the radiographic evaluation of the affected knee.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of Knee Society Score (KSS) equal or greater than "Good" (score ≥ 70) 2 years after surgery | 2 years after surgery
  0-100 scale. Scores rating from 80 to 100 are considered excellent, between 70 and 79 good, between 60 and 69 fair, and less than 60 poor

SECONDARY OUTCOMES:
Changes in Range of Motion over time up to 2 years after surgery | From preoperative to 2 years after surgery
Changes in Oxford Knee Score (OKS) over time up to 2 years after surgery. | From preoperative to 2 years after surgery
  Overall score from 0 to 48, with 48 being the best outcome
Changes in Forgotten Joint Score (FJS) over time up to 2 years after surgery. | From preoperative to 2 years after surgery
  Overall score from 0 to 100, with 100 being the best outcome
Changes in Visual Analogue Scale (VAS) Pain over time up to 2 years after surgery. | From preoperative to 2 years after surgery
  100 mm line, with 0 mm being best outcome (no pain) and 100 mm worst outcome (very severe pain)
Radiographic implant evaluation and stability assessment from postoperative (baseline) over time up to 2 years after surgery | From preoperative to 2 years after surgery
  The treated knee is analyzed postoperatively based on anteroposterior and lateral x-rays view of the knee. The following parametner are evaluated:
  * Presence of radiolucent lines
  * Presence of osteolysis
  * Presence of loosening
  * Presence of heterotopic ossification
  * Presence of periprosthetic fractures
Survival rate (Kaplan-Meier) at 2 years after surgery | From preoperative to 2 years after surgery
Incidence, type and severity of Adverse Device Effects (ADE) and Serious Adverse Device Effects (SADE) up to 2 years follow up | From preoperative to 2 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Tripodo, Principal Investigator — Casa di Cura San Camillo Hospital
Locations (3):
- Italy (3):
  - Casa di Cura San Camillo Hopital, Forte dei Marmi, Lucca
  - Casa di Cura Carmona, Messina
  - Istituto Clinico Porta Sole, Perugia